CLINICAL TRIAL: NCT04152330
Title: Proposal for Parental Guidance and Early Stimulation in Children With Congenital Heart Disease: Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5553/18
Record Dates: First submitted 2019-06-25; First posted 2019-11-05 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2020-07

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Children developmental; Parents training
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison between intervention and control group (Other): The subjects will be randomized to two groups, intervention group (IG) and control group (CG). Each day GI Parents-Baby receives guidance for 6 weeks of stimulation activities and will be instructed to keep an online execution diary, directly with the researcher of videos and messages via cell phone. "Parents" is understood as a generalist nomenclature and will be considered a parent, mother or principal.
  GC subjects receive standard guidance from the pediatric and pediatric cardiology clinic.
  Interventions: Other: Early stimulation protocol on neuropsychomotor development of children with congenital heart disease

INTERVENTIONS:
Other: Early stimulation protocol on neuropsychomotor development of children with congenital heart disease — A parenting guidance booklet will be prepared. It will contain a specific program of stimulation activities for each stage of development in simple language and with illustrations. Subdivided into 4 areas: Cognition, Language, Large Motor and Fine Motor. The duration will be 6 weeks. Parents will participate in 1 individual face-to-face meeting, where they will receive information and clarification on the application of the booklet and will have a mobile communication channel to answer questions throughout the process. Parents will be instructed on the capabilities and limitations of their babies according to the child's congenital heart disease, as well as what is expected within the typical development for this age group and the importance of early stimulation activities in each child in 4 areas of development.

SUMMARY:
Problem: With the increased survival rate of children with congenital heart disease, other health problems, in addition to the clinic, have emerged, such as the risks of developmental delay to which these children are exposed. There is a need for low-cost intervention studies that seek to minimize these risks.

Objective: To evaluate the effect of an early stimulation program using parents as vectors of intervention, on the neurodevelopment of children with CHD Methodology: Randomized clinical trial, conducted with 44 dyads of parents-babies with CH considered as medium and high risk for developmental delays according to the guidelines of the American Heart Association (2012). The study will consist of two groups G1 (Intervention) and G2 (controls). G1 parents will receive guidance for 6 weeks of stimulation activities and will be instructed to keep an online execution diary, direct with the researcher through videos, and messages via cell phone. G2 parents will receive the standard guidelines currently used in pediatric cardiology clinics. Children from both groups will be assessed at the beginning and end of the 6 weeks by the Bayley Baby and Toddler Development Scales (3rd Edition). A questionnaire on the applicability of the protocol will be administered to the parents of the intervention group Expected results: Better neuropsychomotor performance in children after applying the early stimulation protocol.

Perspectives: Create a body of information that can serve as a basis for the formulation of policies for intervention and surveillance of the development of this population.

ELIGIBILITY:
Inclusion criteria:

For babies

* Diagnosis of congenital heart disease up to 3 months old.
* Stable clinical condition (with medical clearance to receive the intervention), For parents
* Parents are literate
* Acceptance of the Responsible to participate in the research.
* Have a mobile device capable of sending and receiving messages and videos.

Exclusion criteria:

For babies

* Suspected or diagnosed genetic syndrome;
* Musculoskeletal or neurological malformation associated
* inability to establish a primary caregiver as in the case of baby under state supervision.

for parents

* Illiteracy
* Presence of deafness, blindness or physical disability, when another family member cannot be responsible for the application of the protocol.

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Difference between groups | 6 moths
  Early intervention prevents developmental delays in children with congenital heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Lucchese, Doutora, Principal Investigator — Instituto de cardiologia de porto alegre
Locations (1):
- Instituto de cardiologia de porto alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No